CLINICAL TRIAL: NCT00806416
Title: A 2-Part, Open-Label, Randomized, Crossover Study to Evaluate the Bioequivalence of the 70 mg Alendronate/2800 IU Vitamin D3 Final Market Combination Tablet to a 70 mg Alendronate Marketed Tablet, and the Relative Bioavailability of Vitamin D3
Brief Title: A Study of the Bioequivalence of 70 mg Alendronate and 70 mg Alendronate in Combination With 2800 IU Vitamin D
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0217A-226; 2008_596
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Results first posted 2010-02-12 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Alendronate; Cholecalciferol; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1 (Experimental): alendronate/vitamin D combination then alendronate
  Interventions: Drug: alendronate sodium (+) cholecalciferol; Drug: Comparator: alendronate
- Sequence 2 (Experimental): alendronate then alendronate/vitamin D combination
  Interventions: Drug: alendronate sodium (+) cholecalciferol; Drug: Comparator: alendronate
- Sequence 3 (Experimental): alendronate/vitamin D combination then vitamin D
  Interventions: Drug: alendronate sodium (+) cholecalciferol; Dietary Supplement: Comparator: cholecalciferol (Vitamin D)
- Sequence 4 (Experimental): vitamin D then alendronate/vitamin D combination
  Interventions: Drug: alendronate sodium (+) cholecalciferol; Dietary Supplement: Comparator: cholecalciferol (Vitamin D)

INTERVENTIONS:
Drug: alendronate sodium (+) cholecalciferol — A single dose tablet of 70 mg alendronate/2800 IU (international unit) vitamin D in one treatment period of each sequence. There will be a 12 day interval between each treatment period.
Drug: Comparator: alendronate — A single dose table of 70 mg alendronate in one treatment period of each sequence. There will be a 12 day interval between each treatment period.
  Arms: Sequence 1; Sequence 2
Dietary Supplement: Comparator: cholecalciferol (Vitamin D) — A single dose tablet of 2800 IU vitamin D in one treatment period of each sequence. There will be a 12 day interval between each treatment period.
  Arms: Sequence 3; Sequence 4

SUMMARY:
This study will evaluate the bioequivalence of alendronate in combination with vitamin D (cholecalciferol) compared to alendronate alone and the bioequivalence of vitamin D in combination with alendronate compared to vitamin D alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or nonpregnant female age 18 to 65 years
* Female of childbearing potential on appropriate method of contraception and not nursing
* BMI (body mass index) less than or equal to 30 kg/m2
* Subject is in good health
* Willing to limit direct sunlight and apply sunscreen if in the sun more than 1 hour

Exclusion Criteria:

* mental or legal incapacitation
* received bisphosphonate treatment within 3 months of screening
* unable to sit or stand upright for at least 2 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2003-05; Primary Completion 2003-08 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Denker AE, Lazarus N, Porras A, Ramakrishnan R, Constanzer M, Scott BB, Chavez-Eng C, Woolf E, Maganti L, Larson P, Gottesdiener K, Wagner JA. Bioavailability of alendronate and vitamin D(3) in an alendronate/vitamin D(3) combination tablet. J Clin Pharmacol. 2011 Oct;51(10):1439-48. doi: 10.1177/0091270010382010. Epub 2010 Dec 8. PMID 21148044

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the following clinical research organizations: Thomas Jefferson University, Division of Clinical Pharmacology, Philadelphia, PA; Clinical Pharmacology Associates, Miami, FL; and Northwest Kinetics, Tacoma, WA, between May 2003 and July 2003.
Pre-assignment Details: A total of 244 participants were enrolled in the study (214 participants were enrolled in Part I and 30 participants were enrolled in Part II).
Groups:
- Alendronate/Vitamin D Combination Then Alendronate: 70 mg alendronate/2800-IU (international unit) vitamin D3 (cholecalciferol) combination tablet; 70 mg alendronate tablet
- Alendronate Then Alendronate/Vitamin D Combination: 70 mg alendronate tablet; 70 mg alendronate/2800-IU vitamind D3 comination tablet
- Alendronate/Vitamin D Combination Then Vitamin D: 70 mg alendronate/2800-IU vitamind D3 combination tablet; 2800-IU vitamin D3 tablet
- Vitamin D Then Alendronate/Vitamin D Combination: 2800-IU vitamin D3 tablet; 70 mg alendronate/2800-IU vitamin D3 comination tablet
Period: Period 1 - Part I
Arm/Group | Alendronate/Vitamin D Combination Then Alendronate | Alendronate Then Alendronate/Vitamin D Combination | Alendronate/Vitamin D Combination Then Vitamin D | Vitamin D Then Alendronate/Vitamin D Combination
Started | 107 | 107 | 0 | 0
Completed | 104 | 103 | 0 | 0
Not Completed | 3 | 4 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 0
Period: Period 2 - Part I
Arm/Group | Alendronate/Vitamin D Combination Then Alendronate | Alendronate Then Alendronate/Vitamin D Combination | Alendronate/Vitamin D Combination Then Vitamin D | Vitamin D Then Alendronate/Vitamin D Combination
Started | 104 | 103 | 0 | 0
Completed | 104 | 103 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Period 1 - Part II
Arm/Group | Alendronate/Vitamin D Combination Then Alendronate | Alendronate Then Alendronate/Vitamin D Combination | Alendronate/Vitamin D Combination Then Vitamin D | Vitamin D Then Alendronate/Vitamin D Combination
Started | 0 | 0 | 14 | 16
Completed | 0 | 0 | 14 | 14
Not Completed | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Period: Period 2 - Part II
Arm/Group | Alendronate/Vitamin D Combination Then Alendronate | Alendronate Then Alendronate/Vitamin D Combination | Alendronate/Vitamin D Combination Then Vitamin D | Vitamin D Then Alendronate/Vitamin D Combination
Started | 0 | 0 | 14 | 14
Completed | 0 | 0 | 14 | 14
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part I: 70 mg alendronate/2800-IU vitamin D3 combination tablet; 70 mg alendronate tablet
- Part II: 2800-IU vitamin D3 tablet; 70 mg alendronate/2800-IU vitamin D3 comination tablet
- Total: Total of all reporting groups
Arm/Group | Part I | Part II | Total
Number analyzed (Participants) | 214 | 30 | 244
Age, Continuous [Mean (Full Range); unit: years] | 41.6 [18 to 65] | 35.2 [19 to 54] | 40.8 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 14 | 133
  Male | 95 | 16 | 111
Height [Mean (Full Range); unit: Centimeters] | 167.2 [144.8 to 190.5] | 170.4 [156.2 to 190.5] | 167.5 [144.8 to 190.5]
Weight [Mean (Full Range); unit: Kilograms] | 72.8 [48.0 to 105.4] | 71.2 [49.9 to 98.4] | 72.6 [48.0 to 105.4]

OUTCOME MEASURES:

1. Primary Outcome: Part 1: The Total Urinary Excretion of Alendronate With Alendronate/Vitamin D Combination Tablet Relative to Alendronate Tablet
Description: Urinary excretion of alendronate was determined over a 36-hour period following single-dose administration of a 70 mg alendronate/2800-IU vitamin D3 combination tablet or 70 mg alendronate alone tablet. Urine for each treatment period was collected at -2 to 0 hours predose, 0 to 8, 8 to 24, and 24 to 36 hours postdose.
Time Frame: On Day 1 across the 36-hour urinary collection period (Periods 1 and 2).
Population: Two hundred-seven (207) subjects (excluding 7 that were enrolled but did not complete both study periods) were included in the statistical analysis.
Measure: Least Squares Mean (Standard Deviation); unit: micrograms (μg)
Groups:
- Alendronate/Vitamin D Combination: 70 mg alendronate/2800-IU vitamin D3 combination tablet
- Alendronate: 70 mg alendronate tablet
Arm/Group | Alendronate/Vitamin D Combination | Alendronate
Number analyzed (Participants) | 207 | 207
micrograms (μg) | 197.5 (329.1) | 191.9 (522.2)
Statistical Analysis 1: Comparison: Alendronate/Vitamin D Combination vs Alendronate; If the true geometric mean ratio (GMR) for total urinary excretion of alendronate of 70 mg alendronate/vitamin D3 combination tablet with respect to alendronate alone is 1.00 then a sample size =208 provided 99% probability of yielding a 90% CI for the total urinary excretion GMR within the interval of [0.80, 1.25]. These calculations were based on the observed-pooled within-subject standard deviation (log scale) of 0.521 obtained from earlier Phase 1 studies; Test type: Non-Inferiority or Equivalence — Administration of a 70 mg alendronate/2800 IU vitamin D3 final market combination tablet and the 70 mg alendronate market tablet, the GMR of the combination tablet/alendronate only tablet are contained within [0.80,1.25]; Least square mean ratio = 1.03, 90% CI [0.91 to 1.17]

2. Primary Outcome: Part II : The Pharmacokinetic Parameters AUC0-120 hr of Vitamin D in Combination Tablet Relative to Vitamin D Tablet
Description: Serum vitamin D3 pharmacokinetic parameter AUC0-120 hr (area under the serum concentration-time curve) after treatment on Day 1was calculated following single-dose administration of a 70 mg alendronate/2800-IU vitamin D3 combination tablet or 2800-IU vitamin D3 tablet.
  Serum for each treatment period was collected at -24, -18, -12, -6, and 0 hours predose, and 2, 3, 5, 7, 9, 12, 16, 24, 36, 48, 72, 96, and 120 hours postdose.
Time Frame: On Day 1 across the 120-hour plasma collection period (Periods 1 and 2).
Population: Twenty-eight (28) subjects (excluding 2 that were enrolled but did not complete both study periods) were included in the statistical analysis.
Measure: Least Squares Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Vitamin D: 2800-IU vitamin D3 tablet
Arm/Group | Alendronate/Vitamin D Combination | Vitamin D
Number analyzed (Participants) | 28 | 28
ng*hr/mL | 296.4 (375.5) | 337.9 (344.2)
Statistical Analysis 1: Comparison: Alendronate/Vitamin D Combination vs Vitamin D; If the true GMRs for AUC and Cmax for 70 mg alendronate/vitamin D3 combination tablet with respect to 2800 IU vitamin D3 alone were 1.00 then a sample size=28 provided >99% probability of yielding a 90% CI for both AUC(0-120 hr) and Cmax GMRs within the interval of [0.80, 1.25]. The within-subject standard deviation of 0.14 ln ng•hr/mL for AUC(0-120 hr) (ng•hr/mL) and 0.14 ng/mL for Cmax was obtained from another phase 1 study; Test type: Non-Inferiority or Equivalence — Administration of a 70 mg alendronate/2800 IU vitamin D3 final market combination tablet and a tablet containing 2800 IU vitamin D3, the geometric mean ratio (GMR) for AUC0-120 hr and Cmax, corrected for predose concentration, of the combination tablet/2800 IU vitamin D3 only tablet were contained within [0.80,1.25]; Least square mean ratio for AUC0-120 hr = 0.88, 90% CI [0.81 to 0.95]

3. Primary Outcome: Part II : The Pharmacokinetic Parameters Cmax of Vitamin D in Combination Tablet Relative to Vitamin D Tablet
Description: Serum vitamin D3 pharmacokinetic parameter Cmax (maximum concentration observed in serum) after treatmen on Day 1was calculated following single-dose administration of a 70 mg alendronate/2800-IU vitamin D3 combination tablet or 2800-IU vitamin D3 tablet. Serum for each treatment period was collected at -24, -18, -12, -6, and 0 hours predose, and 2, 3, 5, 7, 9, 12, 16, 24, 36, 48, 72, 96, and 120 hours postdose.
Time Frame: On Day 1 across the 120-hour plasma collection period (Periods 1 and 2).
Measure: Least Squares Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alendronate/Vitamin D Combination | Vitamin D
Number analyzed (Participants) | 28 | 28
ng/mL | 5.9 (3.3) | 6.6 (3.1)
Statistical Analysis 1: Comparison: Alendronate/Vitamin D Combination vs Vitamin D; If the true GMR ratios for AUC and Cmax for 70 mg alendronate/vitamin D3 combination tablet with respect to 2800 IU vitamin D3 alone were 1.00 then a sample of N=28 provided >99% probability of yielding a 90% CI for both AUC0-120 hr and Cmax GMRs within the interval of [0.80, 1.25]. The within-subject standard deviation of 0.14 ln ng•hr/mL for AUC0-120 hr (ng•hr/mL) and 0.14 ng/mL for Cmax was obtained from another phase 1 study; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; least-squares mean for Cmax = 0.89, 90% CI [0.84 to 0.95]

ADVERSE EVENTS:
Description: 214 subjects were enrolled in Part I of the study & 30 subjects were enrolled in Part II. All 214 subjects in the Alendronate arm & 210 subjects from Part I and 30 subjects from Part II in the Alendronate/Vitamin D Combination are included in the analysis for safety. The 30 Vitamin D arm subjects that were enrolled in Part II are included.
Arm/Group | Alendronate/Vitamin D Combination | Alendronate | Vitamin D
Serious Adverse Events (participants affected / at risk) | 0/240 | 0/214 | 0/30
Other Adverse Events (participants affected / at risk) | 55/240 | 39/214 | 9/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alendronate/Vitamin D Combination (N=240) | Alendronate (N=214) | Vitamin D (N=30)
Conjunctivitis (Eye disorders) | 1 | 0 | 1
Keratoconjunctivitis Sicca (Eye disorders) | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 3 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 6 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 4 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0
Intestinal Functional Disorder (Gastrointestinal disorders) | 1 | 0 | 0
Loose Stools (Gastrointestinal disorders) | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 4 | 4 | 1
Retching (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 3 | 0
Chest Pain (General disorders) | 2 | 2 | 0
Pain (General disorders) | 3 | 1 | 0
Rigors (General disorders) | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 2 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Soft Tissue Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Body Temperature Increased (Investigations) | 0 | 1 | 0
Haemoglobin Decreased (Investigations) | 1 | 0 | 1
White Blood Cells Urine Positive (Investigations) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 3 | 1 | 0
Headache (Nervous system disorders) | 30 | 20 | 3
Somnolence (Nervous system disorders) | 1 | 1 | 0
Haematospermia (Reproductive system and breast disorders) | 1 | 0 | 0
Menstruation Irregular (Reproductive system and breast disorders) | 1 | 0 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hot Flush (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.